CLINICAL TRIAL: NCT01279980
Title: Continuous Wound Infiltration With Local Anaesthetic vs. Epidurals in an Enhanced Recovery Protocol: A Randomised Controlled Trial
Brief Title: Clinical Trial Comparing Epidurals and Local Anaesthetic Wound Catheters in Patients Having Bowel Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scarborough General Hospital (Other)
Responsible Party: Miss Eleanor Richards, Scarborough General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10/H1308/63
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: Pain
Keywords: ERAS; Local anaesthetic wound catheter; Painbuster; Epidural; colorectal surgery; enhanced recovery program
MeSH Terms: conditions — Pain | interventions — Injections, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epidural (Active Comparator): Subjects will have an epidural catheter placed to provide postoperative pain relief. This is standard care for those undergoing an enhanced recovery program.
  Interventions: Other: Epidural
- Painbuster (Active Comparator): Subjects will have a local anaesthetic wound catheter inserted into the wound at time of surgery rather than an epidural for the provision of postoperative pain relief.
  Interventions: Other: Local anaesthetic wound catheter

INTERVENTIONS:
Other: Epidural — Epidural analgesia inserted prior to surgery to stay in until at least the second postoperative day
  Arms: Epidural
Other: Local anaesthetic wound catheter — The catheter will be used to infuse the wound with local anaesthetic for 48 hours post op.
  Other Names: Painbuster(registered trademark)
  Arms: Painbuster

SUMMARY:
The purpose of this study is to find out whether the use of Painbuster® (a local anaesthetic wound catheter) can be used instead of epidurals for patients having bowel surgery in an enhanced recovery programme. The investigators want to find out whether or not using this device means people need to stay in hospital for less time after surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are undergoing either laparoscopic or open colorectal resection will be considered eligible for the study.

Exclusion Criteria:

* Patients under 18 years of age
* Pregnant females
* Patients undergoing an abdominoperineal resection
* Patients unable to understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | determined on discharge from hospital
  Length of stay will be measured in days for each group.This will be determined by a set of predefined discharge criteria.

SECONDARY OUTCOMES:
Postoperative complications | Whilst an inpatient
  All complications in the postoperative period will be recorded. Particular emphasis will be given to:
  * Wound infection: this will be defined as clinical evidence of purulent discharge and erythema accompanied by microbiological (culture of microorganisms) and haematological evidence (raised white cell count)
  * Cardiac failure: This will be defined as the presence of clinical signs of fluid overload accompanied by radiological features on a chest X-Ray.
  * Complications related to epidural/spinal
  * Adequacy of deep vein thrombosis prophylaxis
Episodes of hypotension in the postoperative period | whilst an inpatient
  This will be defined as a systolic blood pressure of less than 90 mmHg
Postoperative pain | as an inpatient
  This will be assessed objectively using the visual analogue scale for pain. Measurements will be taken twice a day for as long as the epidural catheter or Painbuster® is in situ. Pain scores will be measured at rest and on coughing.
Amount of postoperative IV fluid administered | as an inpatient
  This will be documented on each postoperative day.
Body composition | Tests will be performed daily until the epidural or Painbuster® has been removed.
  Body composition (Fat Mass, Fat Free Mass, Extracellular Fluid Volume, Intracellular Fluid Volume, and Total Body Water) will be determined using a bioelectrical impedence analysis (BIA) machine, specifically the "Bodystat" machine.
Postoperative analgesic requirement | As an inpatient
  The total quantity and type (opiate or non-opiate) of all analgesics administered during the period when epidurals or Painbuster® was in situ will be recorded.
Postoperative stress response | As an inpatient
  This will be assessed using:
  SIRS criteria C reactive protein Indirect calorimetry on alternate days at a fixed time.
Anaesthetic time required | On the day of operation
  he time taken in minutes for insertion of epidural or wound catheter will be recorded in each group.
Postoperative mobility | as an inpatient
  Postoperative mobility will be assessed as time until sit to stand aided and unaided, duration of time spent out of bed on each postoperative day and maximum walking distance with assistance on a daily basis. In addition, assessment of mobilisation will be carried out by the physiotherapists who will record this in patient notes.
  All patients will be given pedometer to wear which will count the number of steps taken. Pedometer readings will be taken twice a day. Pedometers have been previously validated as an objective measurement of mobility.
Day of return of gut function | As an inpatient
  Return of gut function will be defined by the tolerance of >/= 80% of the prescribed nutritional requirement. This will be assessed by a dietician.

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor R Richards, BM Medicine, Principal Investigator — Scarborough General Hospital
Locations (1):
- Scarborough General Hospital, Scarborough, North Yorkshire, United Kingdom